CLINICAL TRIAL: NCT00818051
Title: Randomized Trial Testing Dose Escalated Intensity Modulated Radiotherapy for Women Treated by Breast Conservation Surgery and Appropriate Systemic Therapy for Early Breast Cancer
Brief Title: Radiation Therapy in Treating Women Who Have Undergone Breast Conservation Surgery and Systemic Therapy for Early Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000629770; ICR-IMPORT-HIGH; ICR-CTSU/2007/10013; ISRCTN47437448; EU-20897
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

ARMS (3):
- Arm I (control) (Active Comparator): Patients undergo sequential boost dose intensity-modulated radiotherapy (IMRT) 5 days a week for 4.6 weeks (23 fractions; 56 Gy).
  Interventions: Radiation: intensity-modulated radiation therapy
- Arm II (Experimental): Patients undergo concurrent boost dose IMRT 5 days a week for 3 weeks (15 fractions; 48 Gy).
  Interventions: Radiation: intensity-modulated radiation therapy
- Arm III (Experimental): Patients undergo concurrent boost dose IMRT 5 days a week for 3 weeks (15 fractions; 53 Gy).
  Interventions: Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Radiation: intensity-modulated radiation therapy — Given as 48, 53, or 56 Gy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy, such as intensity-modulated radiation therapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. It is not yet known which radiation therapy schedule is more effective in treating breast cancer.

PURPOSE: This randomized phase III trial is studying three different radiation therapy schedules to compare how well they work in treating women who have undergone breast conservation surgery and systemic therapy for early breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test dose-escalated intensity-modulated radiotherapy after breast conservation surgery in women with early breast cancer who are at higher than average risk for local recurrence.

OUTLINE: This is a multicenter study. Patients are stratified according to center. Patients are randomized to 1 of 3 treatment arms.

* Arm I (control): Patients undergo sequential boost dose intensity-modulated radiotherapy (IMRT) 5 days a week for 4.6 weeks (23 fractions; 56 Gy).
* Arm II: Patients undergo concurrent boost dose IMRT 5 days a week for 3 weeks (15 fractions; 48 Gy).
* Arm III: Patients undergo concurrent boost dose IMRT 5 days a week for 3 weeks (15 fractions; 53 Gy).

Quality-of-life questionnaires are administered at baseline, 6 months, and at 1, 3, and 5 years. Photograph assessments of the breasts are taken at baseline and at 3 and 5 years. Blood samples are collected at baseline and periodically thereafter. Tissue samples are also collected from primary tumor, including new primary tumor in either breast, and recurrent tumor.

After completion of study treatment, patients are followed annually for 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Resectable, unilateral disease
  * T1-3, N0-1, M0 disease
* Has undergone prior breast conservation surgery with complete microscopic resection AND received appropriate systemic therapy for early breast cancer
* Requires a tumor bed boost plus whole breast radiotherapy as indicated by ≥ 1 of the following:

  * Age 18-49 years
  * Tumor size > 2.0 cm after primary surgery (maximum microscopic diameter of invasive component)
  * Tumor of any size treated by primary medical therapy
  * Grade III disease
  * Minimum microscopic margin of noncancerous tissue < 5 mm (excluding deep margin if at deep fascia)
  * Lymphovascular invasion
  * Axillary node positive
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* No prior malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior mastectomy
* No concurrent chemotherapy except primary or sequential chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2008-08

PRIMARY OUTCOMES:
Palpable induration inside the boost volume of the irradiated breast

SECONDARY OUTCOMES:
Other late adverse effects in normal tissue as measured by clinical and photographic assessments and patient self-assessments (quality-of-life questionnaires)
Local tumor control
Location of tumor relapse in breast
Contralateral primary tumors
Regional and distant metastases
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom